CLINICAL TRIAL: NCT03872973
Title: The Effect of Visual Input on Balance, Neural Feedback, Function and Running Mechanics in Athletes With Chronic Ankle Instability
Brief Title: The Effect of Visual Input in Athletes With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Serkan Uzlaşır, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018.14.163
Record Dates: First submitted 2019-03-06; First posted 2019-03-13 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Ankle Injuries
Keywords: balance; chronic ankle instability; function; running
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training Group (Experimental): Neuromuscular training will be performed in this group for 6 weeks.
  Interventions: Other: Neuromuscular Training
- Strobe Group (Experimental): This group will perform neuromuscular training for 6 weeks with a strobe glasses.
  Interventions: Other: Neuromuscular Training; Other: Strobe Glasses
- Control Group (No Intervention): This group will not perform any neuromuscular training program.

INTERVENTIONS:
Other: Neuromuscular Training — The experimental group will perform neuromuscular exercise for 6 weeks.
  The other experimental group will perform neuromuscular exercises with strobe glasses.
  Arms: Strobe Group; Training Group
Other: Strobe Glasses — Stroboscopic glasses, which is characterized by intermittent vision obstruction, is a clinical tool that allows clinicians to examine sensory feedback in a progressive manner without fully seeing visual information.
  Arms: Strobe Group

SUMMARY:
The aim of this study is to investigate the effect of neuromuscular training on balance by using stroboscopic glasses in athletes with chronic ankle instability.

DETAILED DESCRIPTION:
Lateral ankle sprain (LAB) is one of the most common musculoskeletal injuries of 15% of all injuries reported in all sports.Chronic ankle instability (CAI) is characterized by life-long persistent symptoms in 40% of people with recurrent LAB sprain.

It has been reported that there is a change in sensorimotor function in the activity of individuals with CAI, and they are more dependent on visual information in balance parameters on one leg.While the somatosensory input was clinically feasible; The obstruction of the visual input has been limited in two ways, the eyes being fully open or fully enclosed.However, this changing dynamic has provided a means for the prevention of visual input during more sporty maneuvers, to directly reach compensatory neuroplastic sequelae after injury and to function in a functional way to train the neuromuscular system.This technological innovation makes this possible by reducing the visual input without completely eliminating it.This innovation, called stroboscopic goggles technology, provides a mechanism to disrupt to any degree between eyes closed and open in the visual system.

Stroboscopic vision, characterized by intermittent vision obstruction, can be a clinical tool that allows clinicians to study sensory feedback in a progressive manner without fully seeing visual information. So use stroboscopic goggles to prevent visual information, you can improve the functionality by emphasizing the somatosensor information.In particular, visual manipulations can significantly influence the healthy adult electrocortical dynamics and balance control by triggering the contradiction between visual adult, vestibular and proprioceptive inputs.

The aim of this study, which was planned for this purpose, will be to evaluate the effects of neuromuscular exercises performed on stroboscopic environment on equilibrium, neural feedback and running mechanics.

ELIGIBILITY:
Inclusion Criteria:

1. To have at least 5 years active athletes in any sports branch.
2. The first sprain history of individuals should be inflammatory symptoms (pain, swelling) at least 1 year before the study,
3. Individuals should have unilateral ankle sprain,
4. The newest sprain must have occurred 3 months before or after the date of commencement,
5. Individuals must have at least 2 times a feeling of instability within 6 months,
6. Individuals should not have any ankle fractures in the past
7. Individuals should have undergone no surgical procedure to affect the sensorimotor function in the lower extremity.
8. IDFAI (Identification of Functional Ankle Instability Questionare) score is above 11,
9. FAAM (Foot and Ankle Ability Measure) score less than 90%,
10. FAAM-S (Foot and Ankle Ability Measure Sport Scale) score should be less than 80%.

Exclusion Criteria:

1. Individuals who are not active athletes for at least 5 years in any sports branch.
2. First sprain history of individuals with inflammatory symptoms (pain, swelling) at least 1 year before the study.
3. The absence of unilateral ankle sprain by individuals.
4. The most recent buckling is that it did not take place 3 months before or after the date of commencement.
5. Individuals should not have a feeling of instability for at least 2 times within 6 months.
6. People experience ankle fractures in the past.
7. Individuals have undergone surgery to affect the sensorimotor function in the lower extremity.
8. IDFAI (Identification of Functional Ankle Questionability) score not more than 11.
9. FAAM (Foot and Ankle Ability Measure) score not less than 90%. FAAM-S (Foot and Ankle Ability Measure Sport Scale) score not less than 80%.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
FAAM (Foot and Ankle Ability Measure), | 8 weeks
  Pre-test evaluation will be done. After the end of neuromuscular training for 6 weeks, the final test will be evaluated. This value will be saved as %.
Ankle ROM | 2 weeks
  The two bars of Optojump are placed on the treadmill with a speed of 3.5m / sec and the foot strokes, imbalance and heel strokes will be recorded and the normal joint movements of the ankle with the Myo-motion device will be recorded.
Balance | 2 weeks
  Static and dynamic balances of athletes before and after neuromuscular training will be evaluated. Center of pressure area (COP) foot pressure point shall be evaluated in mm. And İt is defined as a measure indicative of the time and/or distance a subject spent away from a central point.
EEG (Electroencephalography) | 2 weeks
  The theta and beta waveform of EEG values of people will be measured during the static and dynamic balance evaluation.
FAAM-S (Foot and Ankle Ability Measure Sport Scale) | 8 weeks
  Pre-test evaluation will be done. After the end of neuromuscular training for 6 weeks, the final test will be evaluated. The Sports subscale is scored the same as FAAM (Foot and Ankle Ability Measure) 4 being 'no difficulty at all' to 0 being 'unable to do'. The score on each item are added together to get the item score total. The number of items with a response is multiplied by 4 to get the highest potential score. If the subject answers all 8 items the highest potential score is 32, if one item is not answered the highest potential score is 28, if two are not answered the highest potential score is 24, etc. The item score total is divided by the highest potential score. This value is multiplied by 100 to get a percentage. A higher score represents a higher level of physical function.
BMI (Body Mass Index) | 2 weeks
  Body mass index will be calculated before neuromuscular training. It will be evaluated in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan UZLAŞIR, Study Director — Nevşehir Hacı Bektaş Veli University Sports Science Laboratory
Locations (1):
- Serkan UZLAŞIR, Nevşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No